CLINICAL TRIAL: NCT04314817
Title: Adverse Events Related to Treatments Used Against Coronavirus Disease 2019
Acronym: CovidTox
Status: Completed | Type: Observational
Sponsor: Groupe Hospitalier Pitie-Salpetriere (Other)
Collaborators: CMC Ambroise Paré (Other)
Responsible Party: Principal Investigator, Lee S Nguyen, Principal Investigator, Groupe Hospitalier Pitie-Salpetriere
Other Study IDs: CIC1421-20-04
Record Dates: First submitted 2020-03-17; First posted 2020-03-19 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Coronavirus; Iatrogenic Disease; Acute Kidney Injury; ARDS, Human
MeSH Terms: conditions — Coronavirus Infections; Iatrogenic Disease; Acute Kidney Injury; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients treated for Covid-19
  Interventions: Drug: Any drug used to treat Covid-19

INTERVENTIONS:
Drug: Any drug used to treat Covid-19 — lopinavir/ritonavir, remdesivir, interferon beta-1a, chloroquine and/or azithromycin. This list may be amended at a further date.

SUMMARY:
The outbreak of Covid-19 started several clinical trials and treatment experiments all over the world in the first months of 2020. This study investigates reports of adverse events related to used molecules, including but not limited to protease inhibitors (lopinavir/ritonavir), chloroquine, azithromycin, remdesivir and interferon beta-1a. Analyses of reports also include the International classification of disease ICD-10 for treatments in the World Health Organization (WHO) global Individual Case Safety Report (ICSR) database (VigiBase).

ELIGIBILITY:
Inclusion Criteria:

* all patients treated for Covid-19

Exclusion Criteria:

* Chronology not compatible between the drug and the toxicity

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients treated with a drug that could be reported in the WHO's pharmacovigilance database and with a plausible indication against Covid-19
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2020-03-17 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Renal failure | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms

SECONDARY OUTCOMES:
Heart failure | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
EKG disturbance | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
Hepatic failure | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
Anemia | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
Leucopenia | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
Vascular disease | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
Toxidermia | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
Osteoarticular adverse event | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
Death | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
Acute respiratory distress syndrome | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms
Pulmonary embolism or pulmonary hypertension | Case reported in the World Health Organization (WHO) database of individual safety case reports to 17/03/2020
  defined by the Medical Dictionary for Regulatory Activities (MeDRA) terms

CONTACTS AND LOCATIONS:
Overall Officials: Joe-Elie Salem, MD, PhD, Study Director — Clinical Investigations Center
Locations (1):
- AP-HP Assistance Publique Hopitaux de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No
No individual data is available per se. They need to be retrieved from the World Health Organization.

REFERENCES:
- [Derived] Jung SY, Kim MS, Li H, Lee KH, Koyanagi A, Solmi M, Kronbichler A, Dragioti E, Tizaoui K, Cargnin S, Terrazzino S, Hong SH, Abou Ghayda R, Kim NK, Chung SK, Jacob L, Salem JE, Yon DK, Lee SW, Kostev K, Kim AY, Jung JW, Choi JY, Shin JS, Park SJ, Choi SW, Ban K, Moon SH, Go YY, Shin JI, Smith L. Cardiovascular events and safety outcomes associated with remdesivir using a World Health Organization international pharmacovigilance database. Clin Transl Sci. 2022 Feb;15(2):501-513. doi: 10.1111/cts.13168. Epub 2021 Oct 31. PMID 34719115